CLINICAL TRIAL: NCT01873924
Title: Clinical and Neuropsychological Investigations in Batten Disease
Status: Recruiting | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Jennifer Vermilion, Assistant Professor, University of Rochester
Other Study IDs: Batten Study
Record Dates: First submitted 2013-05-17; First posted 2013-06-10 (Estimated); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Neuronal Ceroid Lipofuscinosis; Neuronal Ceroid Lipofuscinosis CLN1; Neuronal Ceroid Lipofuscinosis CLN2; Neuronal Ceroid Lipofuscinosis CLN3; Neuronal Ceroid Lipofuscinosis CLN5; Neuronal Ceroid Lipofuscinosis CLN6; Neuronal Ceroid Lipofuscinosis CLN7; Neuronal Ceroid Lipofuscinosis CLN8; Neuronal Ceroid Lipofuscinosis CLN10; Batten Disease
Keywords: Batten disease; NCL; Neuronal Ceroid Lipofuscinosis
MeSH Terms: conditions — Neuronal Ceroid-Lipofuscinoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — whole blood, buccal epithelial cells
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- Batten disease: Individuals with any form of Batten disease (Neuronal Ceroid Lipofuscinosis)

SUMMARY:
This study aims to assess the natural history of Batten disease (Neuronal Ceroid Lipofuscinosis) by obtaining information about the motor, behavioral, and functional capabilities of individuals with Batten disease. This study will also refine and validate the Unified Batten Disease Rating Scale (UBDRS) as a clinical rating instrument for Batten disease.

DETAILED DESCRIPTION:
Batten Disease is an inherited disorder that causes progressive cognitive and behavioral decline in children. There have been no systematic clinical studies of Batten Disease using standardized rating instruments with known inter-rater reliability and validity.

The Batten Study Group developed the Unified Batten Disease Rating Scale (UBDRS), a clinical rating instrument used to assess the motor, behavioral, and functional capabilities of individuals with Batten disease. Using the UBDRS, study investigators will evaluate participants approximately every year to track disease progression. The UBDRS is the primary natural history tool, but the study also includes neuropsychological assessment, adaptive function, quality of life measures, and other measures to assess the impact of Batten Disease. Participants will be examined at the University of Rochester Batten Center, Batten Disease Support and Research Association annual meeting, or remotely via televideo. Information related to racial and ethnic background, medical history, symptoms, medications, and diagnostic testing will be collected.

ELIGIBILITY:
Inclusion Criteria:

* child or adult with any form of Batten disease
* parent or legal guardian of a child or adult with any form of Batten disease

Exclusion Criteria:

- parent or guardian unable or unwilling to provide permission for the affected individual

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals diagnosed with any form of Batten disease and their parents/legal guardians are eligible to take part in this study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2004-08; Primary Completion 2035-08 (Estimated); Study Completion 2035-08 (Estimated)

PRIMARY OUTCOMES:
Unified Batten Disease Rating Scale (UBDRS), assessing the severity and change in physical, seizure, behavioral, and functional aspects of individuals with Batten Disease. | Annual Assessments for up to 20 years
  A quantitative measure of natural history

SECONDARY OUTCOMES:
Cognitive and neurobehavioral functioning of individuals with Batten disease | Annual Assessments for up to 10 years
  A standardized battery of neuropsychological tests and neurobehavioral assessments will be used to measure cognitive skills (e.g., verbal reasoning, attention, memory, language), mood, behavior, adaptive function, and quality of life.
Quantitative assessment of vision and retinal thickness | Annual Assessments for up to 20 years
  Vision and retinal thickness assessments include visual acuity, visual fields, fundus photography to document anatomic extent of disease, fundus autofluorescence to measure lipofuscin accumulation, and optical coherence tomography (OCT) to provide detailed images of retinal structure, measure retinal layers, and measure central macular thickness.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan W Mink, MD PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States